CLINICAL TRIAL: NCT00887419
Title: Pain Coping Skills Training for Spinal Cord Stimulator Implant Candidates
Brief Title: Spinal Cord Stimulator Implant Study
Acronym: SCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000226; NIH R01-NS-053759
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Back Pain
Keywords: chronic back pain; spinal cord stimulator implant
MeSH Terms: conditions — Back Pain | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Coping Skills Training (Experimental): Coping Skills Training in pain management
  Interventions: Behavioral: Coping Skills Training
- Education (Active Comparator): Chronic Pain Education
  Interventions: Behavioral: Education
- Usual Care (No Intervention): Patients receive no study intervention, continue with usual medical care.

INTERVENTIONS:
Behavioral: Coping Skills Training — Patients meet individually with therapist for 6 sessions to learn coping skills for stress management, behavioral activation, and communication.
  Arms: Coping Skills Training
Behavioral: Education — Patients meet individually with a health educator for 6 sessions in a presentation/discussion format to receive basic information on the etiology and treatment of chronic pain.
  Arms: Education

SUMMARY:
This study is for patients who have been approved by their doctors and insurance companies to receive spinal cord stimulator implants.

The goal of this study is to investigate if pain and disability is improved in patients with an implant in combination with coping skills training. These patients are compared with those with an implant that receive chronic education information and those with an implant that are in the control group and receive no additional training or information.

DETAILED DESCRIPTION:
This study tests the hypotheses that a pain coping skills program in combination with an SCS implant can improve short- and long-term outcomes in self-efficacy for coping with chronic pain, physical disability, psychological distress, and pain intensity.

Participants are patients who have been approved by their doctors and insurance companies to receive the spinal cord stimulator trial. After patients have been approved, they can be enrolled in this study. After completing a baseline evaluation, patients are randomized into (1)six individual pain coping skills training sessions(relaxations techniques, communication skills, goal setting), (2) six individual chronic pain education sessions (discussion approach to etiology and treatment of chronic pain and information on spinal cord stimulator implants, or (3) treatment as usual (no study intervention).

Participants are evaluated prior to or shortly after their surgery, at post treatment, at 6 month follow-up and at 12 month follow-up. All participants continue their routine medical care throughout the study.

ELIGIBILITY:
Inclusion Criteria

* daily back pain for 6 months or more
* approved by physician and psychologist for implant
* ability to read and write English
* at least 18 years old

Exclusion Criteria:

* pending litigation
* not approved for implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvements in pain, psychological distress, and physical disability | Pre-intervention, post-intervention, 6 month, and 12 month follow-ups
  Improvements in pain, psychological distress, and physical disability Pre-intervention, post-intervention, 6 month, and 12 month follow-ups

SECONDARY OUTCOMES:
Patients will learn a repertoire of coping skills which can be applied to other challenges in life. | Pre-intervention, post intervention, 6 month, and 12 month follow-ups
  Patients will learn a repertoire of coping skills which can be applied to other challenges in Pre-intervention, post intervention, 6 month, and 12 month follow-upslife.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States